CLINICAL TRIAL: NCT00087854
Title: Dose-Defining Study of a NAT2 Phenotype-Based Dosing Regimen of Intravenous Amonafide L-Malate Administered Weekly in Men With Androgen-Independent Prostate Cancer (AIPC)
Brief Title: Study of Individualized Amonafide to Treat Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xanthus Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001A2-200-US
Record Dates: First submitted 2004-07-14; First posted 2004-07-16 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — xanafide; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Amonafide L-malate (drug)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Amonafide in men with androgen-independent prostate cancer, assigned to individualized doses of Amonafide based on acetylator phenotype information (doses adjusted on individual metabolism).

DETAILED DESCRIPTION:
This is an open-label, Phase I/II, multicenter study of Amonafide in subjects with androgen-independent metastatic prostate cancer.

Amonafide is metabolized by N-acetylation to an active metabolite, N-acetyl-Amonafide. Inter-subject differences in N-acetylation can explain the variability in Amonafide-induced myelosuppression. This dose-defining protocol has been designed to assess safety and efficacy of Amonafide in men with androgen-independent prostate cancer, assigned to individualized doses based on acetylator phenotype information.

The total duration of this study will be approximately 12 - 16 months: approximately 6 - 10 months for enrollment, and approximately 6 months for subject screening, treatment, and follow up per protocol. Subjects will be treated until PSA progression, disease progression, or unacceptable toxicity.

Subjects may continue participation in the study after Cycle 5 at the investigator's discretion if PSA progression, disease progression, or unacceptable toxicities are not reported. If a subject fulfills a criterion of PSA progression or disease progression, yet in the opinion of the investigator, the subject appears to be deriving clinical benefit from the study medication, a request may be made to the Xanthus medical monitor to allow that subject to continue study participation on a compassionate basis.

A follow-up evaluation for all subjects will be done 30 - 35 days after receiving the last dose of Amonafide. Subjects will be contacted every 3 months for survival after completion of the active phase of the study, until death.

PSA response will be reported for all subjects receiving Amonafide treatment. PSA levels will be measured at Screening and once per treatment cycle thereafter (at Day 1 of each cycle). A PSA responder will be defined as a subject experiencing a 50% decrease in PSA level, confirmed four or more weeks later, with no demonstration of clinical or radiographic evidence of disease progression prior to the second PSA measurement. Duration PSA response and time to PSA progression will also be reported.

In addition to PSA endpoints, traditional response criteria such as overall tumor response rate (complete + partial tumor response), duration of tumor response, and time to tumor progression will be captured for all subjects with measurable lesions. All complete and partial responses must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are met.

Subsequently, in order to evaluate safety, all subjects will be assessed for signs of adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3 dated June 10, 2003.

All serious adverse events (SAEs) and grade ¾ toxicities will be reviewed by the Sponsor's medical monitor. Appropriate action may be taken to terminate or put the study on hold if warranted by unanticipated toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years or older;
* Metastatic androgen-independent prostate cancer with evidence of progression;
* Zero or one prior course of chemotherapy for metastatic disease;
* Up to two prior courses of non-cytotoxic therapies for metastatic disease;
* Progressive measurable or assessable disease;
* Evidence of continued elevation of PSA despite antiandrogen withdrawal;
* ECOG Performance Status < 2 with an expected survival of at least 6 months;
* Adequate renal function;
* Adequate hepatic function;
* Adequate hematologic status;
* No other prior malignancy is allowed except for the following: adequately-treated basal cell or squamous cell skin cancer, adequately treated Stage I or II bladder cancer from which the subject is currently in complete remission, or any other cancer from which the subject has been disease free for 5 years;
* Subjects must have recovered from all acute toxicities from prior treatment;
* Screening visit phenotyping procedures must have been completed successfully;
* No blood transfusion within the previous 2 weeks of signature of the informed consent;
* Expected cooperation of the subject for the treatment and follow up must be obtained and documented;
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Clinically significant abnormal hematological parameters other than those defined in the inclusion criteria;
* Clinically significant abnormal biochemical parameters other than those defined in the inclusion criteria;
* Subjects who have been receiving bisphosphonates for less than three months prior to the first Amonafide administration;
* Known history of brain metastases;
* Subjects who are HIV positive;
* Subjects who are hepatitis B surface antigen positive or have previously documented hepatitis C infection;
* Subjects who received treatment with Growth Factors (i.e. G-CSF, GM-CSF) within 2 weeks of the signature of the informed consent form;
* Subjects who had any major surgery within four weeks of first administration of Amonafide;
* Subjects with a history of a psychological illness or condition which may interfere with the subjects ability to understand or comply with the requirements of the study;
* Subjects who received an investigational new drug within 30 days of the first dose of Amonafide;
* Any other known condition, which in the investigator's opinion would not make the subject a good candidate for the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The Primary Objectives of this study are:
To define and validate the safety of a NAT2 pheontypically driven dosing regimen;
To define the pharmacokinetic and pharmacodynamic profile of Amonafide with a weekly intravenous administration schedule.

SECONDARY OUTCOMES:
The Secondary Objectives of this study are:
To determine the efficacy of weekly intravenous Amonafide for all enrolled subjects as defined by PSA response (decrease in PSA of 50% or greater), duration of PSA response, and time to PSA progression;
To determine the overall tumor response (e.g., complete response or partial response), duration of tumor response, and time to tumor progression among subjects with measurable lesions using standard (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Drouin, MD, Study Chair — Xanthus Life Sciences-Medical Monitor; Monique Champagne, BPharm, MSc, Study Director — Xanthus Pharmaceuticals, Inc.; Mario Eisenberger, MD, Principal Investigator — Johns Hopkins University Hospital
Locations (8):
- United States (8):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Cancer Center at John Hopkins, Baltimore, Maryland
  - Barnard Cancer Center, St Louis, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Herbert Irving Cancer Center, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington